CLINICAL TRIAL: NCT01776242
Title: Back Pain Outcomes Using Longitudinal Data (BOLD) Registry and Repository
Brief Title: Back Pain Outcomes Using Longitudinal Data (BOLD)
Acronym: BOLD
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); Harvard Vanguard Medical Associates (Other); Henry Ford Health System (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey G. Jarvik, MD, MPH, Professor, University of Washington
Other Study IDs: 39009-EA; 101H5019222-01 (Other: ID)
Record Dates: First submitted 2012-06-13; First posted 2013-01-28 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
Keywords: low back pain; elderly; back pain; lumbar pain; over 65
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall objective of BOLD is to establish a large, community-based registry (at least 5000 subjects) of patients aged 65 years and older presenting with new episodes of healthcare visits for back pain. BOLD's primary aim is to create an infrastructure that allows for the conduct of prospective, controlled studies comparing the effectiveness of diagnostic and treatment strategies for back pain in older adults.

DETAILED DESCRIPTION:
The BOLD registry identifies subjects at the time of a new episode of back pain and captures data in a longitudinal fashion for up to 12 months. The registry captures self-report outcomes data as well as comprehensive utilization data including pharmacy and imaging data through the electronic medical record system. We are applying for additional funding to continue follow-up for up to 4 years from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years
* Primary care visit for low back pain based on ICD9 code
* No prior visits for low back pain within six months

Exclusion Criteria:

* Prior lumbar spine surgery
* Developmental spine deformities
* Inflammatory spondyloarthropathy
* Known spinal malignancy or infection
* Primarily nerve compression-related symptoms
* Serious medical co-morbid condition with life expectancy < 1yr
* No telephone, or planning to move within a year
* Unable to understand English
* Severe mental impairment that would interfere with answering questions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults over age 65
Sampling Method: Probability Sample
Enrollment: 5239 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Roland- Morris Disability Questionnaire | Baseline, 3, 6 and 12 month timepoints
  24-item back pain specific, functional status questionnaire

SECONDARY OUTCOMES:
Change in Pain Numerical Rating Scale (NRS) | Baseline, 3, 6 and 12 month timepoints
  Numerical rating score of pain intensity (0-10 scale)
Change in Brief Pain Inventory | Baseline, 3, 6 and 12 month timepoints
  Pain Interference short form
Change in Patient Expectation Regarding Recovery | Baseline, 3, 6 and 12 month timepoints
  Two questions measuring patient expectations
Change in Patient Health Questionnaire-4 (PHQ-4) | Baseline, 3, 6 and 12 month timepoints
  Depression and Anxiety Scale
Demographics | Baseline
  Demographic information
Change in Euro-Qual-D (EQ-5D) | Baseline, 3, 6 and 12 month timepoints
  Five item general health-related quality of life measure
Change in Falls Assessment | Baseline, 3, 6 and 12 month timepoints
  Two questions regarding frequency of falls and any injuries that resulted
Electronic Medical Record Data | 12 months before and after index visit for back pain
  Imaging, health care utilization, pharmacy, laboratory data extracted from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jarvik, MD, MPH, Principal Investigator — University of Washington; Rick Deyo, MD, MPH, Principal Investigator — Oregon Health and Science University; Janna Friedly, MD, Principal Investigator — University of Washington; Partrick Heagerty, PhD, Principal Investigator — University of Washington; Larry Kessler, ScD, Principal Investigator — University of Washington; Sean Sullivan, PhD, Principal Investigator — University of Washington; Judy Turner, PhD, Principal Investigator — University of Washington; Andy Avins, MD, MPH, Principal Investigator — Kaiser-Permanente of Northern CA; David Nerenz, PhD, Principal Investigator — Henry Ford Health Systems; Srdjan Nedeljkovic, MD, Principal Investigator — Harvard-Vanguard Associates
Locations (3):
- United States (3):
  - Kaiser-Permanente of Northern California, Oakland, California
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan

REFERENCES:
- [Background] Jarvik JG, Comstock BA, Bresnahan BW, Nedeljkovic SS, Nerenz DR, Bauer Z, Avins AL, James K, Turner JA, Heagerty P, Kessler L, Friedly JL, Sullivan SD, Deyo RA. Study protocol: the Back Pain Outcomes using Longitudinal Data (BOLD) registry. BMC Musculoskelet Disord. 2012 May 3;13:64. doi: 10.1186/1471-2474-13-64. PMID 22554166
- [Derived] Jarvik JG, Comstock BA, Heagerty PJ, Turner JA, Sullivan SD, Shi X, Nerenz DR, Nedeljkovic SS, Kessler L, James K, Friedly JL, Bresnahan BW, Bauer Z, Avins AL, Deyo RA. Back pain in seniors: the Back pain Outcomes using Longitudinal Data (BOLD) cohort baseline data. BMC Musculoskelet Disord. 2014 Apr 23;15:134. doi: 10.1186/1471-2474-15-134. PMID 24755158
- See also: Study related information — http://www.backpainproject.org